CLINICAL TRIAL: NCT03003286
Title: Community Based Intervention for Children With ADHD and ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lauren Kenworthy (Other)
Collaborators: Georgetown University (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Lauren Kenworthy, ASSOC CHIEF NEUROPSYCHOLOGY, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-1304-7379
Record Dates: First submitted 2016-11-21; First posted 2016-12-28 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Autism Spectrum Disorder; Attention Deficit-Hyperactivity Disorder; Executive Function
Keywords: Contingency Behavior Management; Flexible; Unstuck; Low Income; Behavior; Coping; Disparity; Problem Solving; Self-Control; impulsive; intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Behavior; Self-Control; Impulsive Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UOT Students and Parents (Experimental): Unstuck and on Target (UOT) provided in the classroom for students at Title 1 schools
  Interventions: Behavioral: Unstuck and on Target (UOT)
- PATSS Students and Parents (Experimental): Parents and Teachers Supporting Students (PATSS) provided in the classroom for students at Title 1 schools
  Interventions: Behavioral: Parents and Teachers Supporting Students (PATSS)

INTERVENTIONS:
Behavioral: Unstuck and on Target (UOT) — Unstuck and on Target (UOT) is a novel and innovative cognitive-behavioral treatment that directly addresses executive functioning and self-regulation deficits in ASD and ADHD. UOT is the first contextually-based EF treatment that targets flexibility, goal-setting and planning through a cognitive-behavioral program centered on self-regulatory scripts that are consistently modeled and reinforced. Parents, teachers, and interventionists will be taught to model and support flexibility across settings. Children will also participate in a peer group intervention setting.
  Arms: UOT Students and Parents
Behavioral: Parents and Teachers Supporting Students (PATSS) — The Contingency Behavior Management (CBM) intervention was developed by the researchers and called Parents and Teachers Supporting Students (PATSS) as a current best practice intervention that was comparable in design to Unstuck and on Target. The goal is to improve child behavioral outcomes by training parents, teachers and interventionists in core principles of behavior management like social learning and behavioral change. Children were also included in small group sessions where they identify their own behavior goals and meaningful reinforcers.
  Arms: PATSS Students and Parents

SUMMARY:
The purpose of this study is to determine whether a new treatment, Unstuck and On Target (UOT), works better, worse, or the same as the best treatment that is available now, Contingency Behavioral Management (CBM), for low income children with Autism Spectrum Disorder (ASD) or Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This project will compare the effectiveness of an innovative community-based cognitive-behavioral Executive Functioning (EF) treatment, Unstuck and On Target (UOT) to the current standard of care, a Contingency Behavioral Management (CBM) program in typically underserved children with ASD or ADHD. Minimizing the impact of EF deficits in these pediatric disorders has broad public health implications, providing the opportunity for improvement in the real-world, long-term outcomes that stakeholders have told the investigators are most important to them: more educational and vocational success, more functional independence and improved Activities of Daily Living skills, and better physical health, with reduced morbidity and mortality. The health disparity that this project addresses is the poorer outcomes and limited treatment choices associated with being a child from a low-income family who also has ADHD or ASD. The research questions are:

1. Which works better for low-income children with ASD, UOT or CBM? Researchers will test the comparative effectiveness of UOT to CBM treatments with low-income children with ASD.
2. Which works better for low-income children with ADHD, UOT or CBM? Researchers will test the comparative effectiveness of UOT to CBM with low-income children with ADHD, a new patient population for UOT.
3. Are the effects of UOT and CBM sustained 9-12 months after treatment? Researchers will assess whether any benefits ascribed to the interventions are maintained about a year after the treatment is completed.

Patients with ASD and ADHD will be recruited for the study from school systems. Half will receive UOT and half will receive CBM. Researchers will recruit interested Title 1 schools that serve very different and diverse populations. Recruitment will occur in several stages. Specifically, school districts will invite individual schools to participate in the trial that have a sufficient number of qualifying children. Interested schools will then contact families and provide information about the study. Interested families will initiate contact with study staff, and individual schools will be entered into the study if they have three or more patients whose families contact study staff. Children will then be scheduled for cognitive/diagnostic evaluation. Recruitment will continue until the target enrollment is reached, and all remaining interested families from enrolled schools are included. Subjects with appropriate assent and consent will be evaluated for eligibility and their school will be randomly assigned to treatment condition.

Cognitive problem-solving abilities, flexibility, planning and organizing, self-regulation, behavior problems, coping skills, and the child's use of non-routine urgent medical care will be measured before and after treatment through a multi-method, multi-informant format, including parent report, blinded classroom observations and blinded direct child measures. Researchers chose measures that have the greatest relevance to functional outcomes and "real world" functioning. Rather than define a single outcome, researchers chose multiple outcome variables, anticipating differential impacts of the treatment modalities on the outcome domains. All of the measures and observations will be gathered at pre- and post-treatment time-points in each treatment year.

Data will be analyzed using a Statistical Package for the Social Sciences (SPSS) v20 and R. A comparison of baseline characteristics will be performed between the treatment groups to assess that the randomization was successful. The characteristics will include demographics as well as the direct child assessments and the behavioral scales. These comparisons will be performed using standard statistical methods, such as t-tests for continuous variables or (exact) chi-squares for dichotomous variables. If any characteristic is unbalanced between treatments, which will be possible with the sample size, secondary analyses will adjust for that characteristic.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit children who are referred by teachers and staff at their school for concerns of flexibility (rather than those who are responding to an advertisement), so that the research will have a "real world" group of children to test the effectiveness of the treatments.
* The recruited participants will have symptoms of ASD or ADHD, will be receiving a combination of mainstream and special education supports, and will qualify to attend pull-out groups in school. All the schools involved are eligible for Title 1 governmental support, indicating that the children are from primarily low-income communities, although the investigators will not be requiring that participant's families themselves meet income cutoffs.
* Potential participants will be evaluated individually and included in the study if they achieve a Full Scale IQ score>70, a verbal mental age>6 years old, and meet DSM-IV-TR criteria for either a Autism Spectrum Disorder or ADHD. IQ and verbal mental age will be measured with the Wechsler Abbreviated Scale of Intelligence, 2nd addition (WASI-2) Verbal, Performance and Full Scale IQ scores (represented as Standard Scores: mean=100; SD=15).
* To evaluate for ASD, research-valid clinical psychologists will administer the Autism Diagnostic Observation Schedule, Second Edition Module 3 (ADOS-2), a gold standard structured play/conversational interview that elicits symptoms of ASD. It produces non-standardized raw scores; higher scores indicate more symptoms. To be included in the study, each child must obtain an ADOS diagnostic algorithm >'ASD' threshold and parents will be asked to complete the Social and Communication Questionnaire (SCQ). In order to include the full autism spectrum, these criteria are relatively inclusive.
* To confirm diagnosis of ADHD, parents will complete the ADHD portion of the MINI-Kid ADHD interview with a trained interviewer, and their child must meet DSM-IV criteria for any Attention Disorder. The researchers will include children who had observable symptoms in two of three settings. As all children will be referred for the study because teachers or staff at their school observed symptoms, the children will have to also meet criteria on the MINI-Kid interview or the trained clinician completing their testing will have to observe notable symptoms, or both, for the child to be included in the study.

Exclusion Criteria:

* Participants will be excluded from the study if they have a diagnosis of bipolar disorder, schizophrenia, or major depression that is currently preventing them from participating in classroom activities.
* Students with anxiety, mild depression, obsessive-compulsive disorder or other problems that do not prevent them from participating in the majority of classroom activities will not be excluded.
* Exclusion will be determined through a two-stage process: First, participants will be screened for comorbid symptoms using the Child Behavior Checklist (CBCL). The CBCL for 6-18 year olds has 118 items that describe specific behavioral and emotional problems. Parents rate their child for how true each item is now or within the past 6 months. One of the PIs, both of whom are licensed psychologists with active clinical practices, will follow-up with a child's teacher if a child scores above a T score of 75 on any of the six DSM-oriented scales other than Attention Deficit/Hyperactivity Problems (Affective Problems; Anxiety Problems; Somatic Problems; Oppositional Defiant Problems; and Conduct Problems).
* The investigators will ask teachers targeted questions to determine to what degree the identified symptoms interfere with the child's ability to participate in the classroom activities or in the treatment group such as "Do you feel that the child can participate in most classroom activities? If not, why? Can they listen to and follow written and verbal instructions? Can they participate in activities with other children when given structure and support?" However, because the school programs involved in this study use an inclusion model, students in these mainstream classrooms are unlikely to meet exclusion criteria.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2014-09-13 (Actual); Primary Completion 2017-08-05 (Actual); Study Completion 2017-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Classroom Observation total raw score at termination of intervention | Baseline, 7-8 months
  15-20 minute classroom observation conducted by a treatment-blind research assistant for every study participant during the academic school day. The following behaviors are coded: Social reciprocity, Following Rules, Transitions, Gets Stuck, Negativity/Overwhelm, and Classroom Participation.

SECONDARY OUTCOMES:
Change in Wechsler Abbreviated Scale of Intelligence--II Block Design- T-score at termination of intervention (post testing) and 1 year later (long-term follow-up) | Baseline, 7-8 months, 19-20 months
  A standardized, normed timed visual construction task that requires efficient nonverbal cognitive problem solving.
Change in Delis-Kaplan Executive Function System - Category Fluency and Switching Accuracy scaled scores at termination of intervention (post testing) and 1 year later (long-term follow-up) | Baseline, 7-8 months,19-20 months
  Standardized, normed, executive function tasks
Change in Executive Function Challenge Task - Flexibility and Planning raw scores at termination of intervention (post testing) and 1 year later (long-term follow-up) | Baseline, 7-8 months, 19-20 months
  Observations of participant behavior when confronted with 3 standardized tasks demanding flexibility and planning are coded on a 3-point scale for each task, and summed across tasks.
Change in Flexibility Interference Questions Questionnaire total raw score at termination of intervention (post testing) and 1 year later (long-term follow-up) | Baseline, 7-8 months, 19-20 months
  A short questionnaire was created by researchers for parents to report how often problems with flexibility interfere with daily adaptive functioning.
Change in Behavior Rating Inventory of Executive Function (BRIEF) - Parent Form - Shift, Plan/Organize, Emotional Control and Global Executive at termination of intervention (post testing) and 1 year later (long-term follow-up)Composite T-scores | Baseline, 7-8 months, 19-20 months
  Parent ratings of participant's executive function-related behaviors
Change in The Child Behavior Checklist (CBCL) - Parent Report Externalizing Behaviors T-scores at termination of intervention (post testing) and 1 year later (long-term follow-up) | Baseline, 7-8 months, 19-20 months
  The CBCL for 6-18 year olds has 118 items that describe specific behavioral and emotional problems, plus two open ended items to describe any additional problems, as well as 20 competence items covering positive, pro-social behaviors. Children's scores are expressed as T scores (mean=50; SD=10) on eight empirically based syndromes scales which are based on factor analyses: Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior. The CBCL will be used to track behavioral change at home as a result of the treatments. Researchers predict that UOT and CBM participants will improve equally on the Aggressive Behavior scale, but that UOT participants will improve more on the CBCL Affective Problems score than CBM participants.
Parent Feedback Form - Acceptability total raw score | 7-8 months
  Parent ratings of acceptability of the intervention
Child Feedback-Acceptability raw score | 7-8 months
  Child ratings of acceptability of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Kenworthy, Ph.D., Principal Investigator — Children's National Health Services; Laura Anthony, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Research Institude, Children's National Heath System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders, 4th Edition, Text Revision. 2000.
- [Background] Clopper CJ, Pearson, ES. The use of the confidence or fiducial limits illustrated in the case of the binomial. Biometrika 26(4): 404-413, 1934.
- [Background] Delis DC, Kaplan E, Kramer JH. Delis Kaplan executive function system (D-KEFS). San Antonio, TX: The Psychological Corporation. 2001.
- [Background] Gioia GA, Isquith PK, Kenworthy L, Barton RM. Profiles of everyday executive function in acquired and developmental disorders. Child Neuropsychol. 2002 Jun;8(2):121-37. doi: 10.1076/chin.8.2.121.8727. PMID 12638065
- [Background] Gioia GA, Isquith PK, Retzlaff PD, Espy KA. Confirmatory factor analysis of the Behavior Rating Inventory of Executive Function (BRIEF) in a clinical sample. Child Neuropsychol. 2002 Dec;8(4):249-57. doi: 10.1076/chin.8.4.249.13513. PMID 12759822
- [Background] Mather N, Wendling BJ. Woodcock-Johnson IV tests of achievement: Examiner manual standard and extended batteries. Rolling Meadows, IL: Houghton Mifflin Harcourt. 2014.
- [Background] Weisz JR, Ugueto AM, Cheron DM, Herren J. Evidence-based youth psychotherapy in the mental health ecosystem. J Clin Child Adolesc Psychol. 2013;42(2):274-86. doi: 10.1080/15374416.2013.764824. Epub 2013 Feb 12. PMID 23402704
- [Background] Wells KC, Pelham WE, Kotkin RA, Hoza B, Abikoff HB, Abramowitz A, Arnold LE, Cantwell DP, Conners CK, Del Carmen R, Elliott G, Greenhill LL, Hechtman L, Hibbs E, Hinshaw SP, Jensen PS, March JS, Swanson JM, Schiller E. Psychosocial treatment strategies in the MTA study: rationale, methods, and critical issues in design and implementation. J Abnorm Child Psychol. 2000 Dec;28(6):483-505. doi: 10.1023/a:1005174913412. PMID 11104313